CLINICAL TRIAL: NCT03553576
Title: The Relationship Between Local Anesthetic Concentration and Volume on Adequate Labor Analgesia With Programmed Intermittent Epidural Bolus
Brief Title: Drug Concentration and Volume on Adequate Labor Analgesia With PIEB
Acronym: CADD2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of continued funding
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Feyce M. Peralta, MD, MS, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00206113
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pain; Anesthesia; Labor Pain
Keywords: Labor pain; Epidural; Obstetric; Labor Analgesia
MeSH Terms: conditions — Pain; Labor Pain

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will be blinded to the assigned randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low volume bolus (Experimental): 6.25 mL administration at 250 ml per hour of a greater density solution (0.1% bupivacaine with fentanyl 2.0 mcg/mL)
  Interventions: Drug: Low volume bolus
- High volume bolus (Experimental): 10 mL administration of a lower density local anesthetic (0.0625% bupivacaine with fentanyl 2.0 mcg/mL).
  Interventions: Drug: High volume bolus

INTERVENTIONS:
Drug: Low volume bolus — Administration of a low-volume bolus (6.25 mL) of greater density solution (0.1% bupivacaine with fentanyl 2.0 mcg/mL) at 250 mL per hour given by CADD pump.
  Arms: Low volume bolus
Drug: High volume bolus — Administration of a high-volume bolus (10 mL) of lower density local anesthetic (0.0625% bupivacaine with fentanyl 2.0 mcg/mL) at 250 mL per hour given by CADD pump.
  Arms: High volume bolus

SUMMARY:
Neuraxial labor analgesia is performed by the administration of a local anesthetic/opioid mixture in the epidural space. The delivery method is a combination of continuous infusion, provider-administered boluses and patient-administered boluses (patient controlled epidural analgesia [PCEA]) via epidural catheter. The anesthetic solution administered through the lumbar epidural catheter must spread cephalad in the epidural space to reach the T10 nerve roots and spinal cord, and must spread caudad to reach the caudal nerve roots in the epidural space.

Epidural infusion pumps capable of delivering PIEB of local anesthetic with PCEA have become commercially available and many studies have attempted to assess the optimal parameter settings (including volume of programmed bolus, bolus interval, rate of bolus administration) to provide superior labor analgesia.

Traditionally higher concentration local anesthetic solutions have been associated with increased motor blockade leading to a higher incidence of instrumental vaginal delivery. Several local anesthetic solutions with varying drug concentrations are available for labor analgesia and are used clinically in the United States. We plan to perform a randomized, controlled, double-blind study to test the hypothesis that patients whose labor analgesia is maintained using PIEB with low-volume bolus (6.25 mL) of a higher local anesthetic concentration solution (0.1% bupivacaine with fentanyl 2.0 mcg/mL) will require less supplemental analgesia (manual provider re-doses) than patients whose PIEB is delivered with a high-volume bolus (10 mL) of lower density local anesthetic solution (0.0625% bupivacaine with fentanyl 2.0 mcg/mL).

The aim of this study is to evaluate the association between bolus volume and concentration of local anesthetic during maintenance of labor analgesia with programmed intermittent epidural bolus (PIEB) analgesia.

The hypothesis of this study is: patients whose labor analgesia is maintained using PIEB with low-volume bolus (6.25 mL) of higher local anesthetic concentration solution (0.1% bupivacaine with fentanyl 2.0 mcg/mL) will have a longer duration of adequate analgesia (time to first manual re-dose request) than patients whose PIEB is delivered with a high-volume bolus (10 mL) of lower concentration local anesthetic solution (0.0625% bupivacaine with fentanyl 2.0 mcg/mL).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Nulliparous parturients
* Present to the labor and delivery unit for an induction of labor or who are in spontaneous labor
* Request neuraxial labor analgesia at ≤5 cm cervical dilation

Exclusion Criteria:

* Patients who are not eligible to receive a combined spinal epidural (CSE) technique with 25 mcg of intrathecal fentanyl
* Non-English speaking
* Failed initiation of CSE analgesia (VAS pain score >10 15 minutes after intrathecal dose)
* Need to have the epidural catheter replaced during labor
* Who deliver within 90 minutes of initiation of labor analgesia
* Require re-dose within 90 minutes of initiation of labor analgesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant female
Enrollment: 146 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feyce Peralta, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Background] Lim Y, Sia AT, Ocampo C. Automated regular boluses for epidural analgesia: a comparison with continuous infusion. Int J Obstet Anesth. 2005 Oct;14(4):305-9. doi: 10.1016/j.ijoa.2005.05.004. PMID 16154735
- [Background] Chua SM, Sia AT. Automated intermittent epidural boluses improve analgesia induced by intrathecal fentanyl during labour. Can J Anaesth. 2004 Jun-Jul;51(6):581-5. doi: 10.1007/BF03018402. PMID 15197122
- [Background] Kaynar AM, Shankar KB. Epidural infusion: continuous or bolus? Anesth Analg. 1999 Aug;89(2):534. doi: 10.1097/00000539-199908000-00063. No abstract available. PMID 10439786
- [Background] Hogan Q. Distribution of solution in the epidural space: examination by cryomicrotome section. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):150-6. doi: 10.1053/rapm.2002.29748. PMID 11915061
- [Background] Comparative Obstetric Mobile Epidural Trial (COMET) Study Group UK. Effect of low-dose mobile versus traditional epidural techniques on mode of delivery: a randomised controlled trial. Lancet. 2001 Jul 7;358(9275):19-23. doi: 10.1016/S0140-6736(00)05251-X. PMID 11454372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited within Prentice Women's Hospital labor and delivery unit. Recruitment period start date was 1/21/2020 and the end date for recruitment was 09/01/2022.
Pre-assignment Details: 146 subjects consented to participate in the study.
Groups:
- Low Volume Bolus 0.1% Bupivacaine: 6.25 mL administration at 250 ml per hour of a greater density solution (0.1% bupivacaine with fentanyl 2.0 mcg/mL)
  Low volume bolus: Administration of a low-volume bolus (6.25 mL) of greater density solution (0.1% bupivacaine with fentanyl 2.0 mcg/mL) at 250 mL per hour given by CADD pump.
- High Volume Bolus .0625% Bupivacaine: 10 mL administration of a lower density local anesthetic (0.0625% bupivacaine with fentanyl 2.0 mcg/mL).
  High volume bolus: Administration of a high-volume bolus (10 mL) of lower density local anesthetic (0.0625% bupivacaine with fentanyl 2.0 mcg/mL) at 250 mL per hour given by CADD pump.
Period: Overall Study
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Started | 73 | 73
Completed | 67 | 62
Not Completed | 6 | 11
Not completed — MD withdrew (pump settings changed d/t interscapular pain) | 1 | 1
Not completed — Unintentional dural puncture during epidural procedure | 0 | 1
Not completed — No cerebral spinal fluid obtained during epidural procedure a straight catheter was used | 0 | 1
Not completed — Fentanyl and or clonidine administered via epidural catheter | 1 | 2
Not completed — First redose of anesthetic by anesthesiologist administered under 90 minutes after catheter placed | 1 | 1
Not completed — Greater than 3 redoses of anesthetic by the anesthesiologist using the epidural catheter | 1 | 0
Not completed — Physician Decision | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine | Total
Number analyzed (Participants) | 67 | 62 | 129
Age, Customized [Mean (Full Range); unit: Years]
  Age | 32.6 [28.5 to 36.7] | 32.9 [28.7 to 37.1] | 32.8 [28.5 to 37.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 129
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 59 | 54 | 113
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 43 | 46 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 67 | 62 | 129
Gestational age [Mean (Full Range); unit: Weeks] | 39.3 [38.3 to 40.3] | 39.6 [38.8 to 40.4] | 39.4 [38.3 to 40.4]
BMI kg/m^2 [Mean (Full Range); unit: kg/m^2] | 29.8 [25.4 to 34.2] | 32.0 [25.8 to 38.2] | 31 [25.4 to 38.2]
Number of times pregnant [Count of Participants; unit: Participants]
  1 time pregnant | 44 | 52 | 96
  2 times pregnant | 20 | 6 | 26
  3 times pregnant or greater | 3 | 4 | 7
Labor type [Count of Participants; unit: Participants]
  Spontaneous labor | 39 | 29 | 68
  Induction of labor | 28 | 33 | 61
Fetal position [Count of Participants; unit: Participants] — The position of the fetus within the uterus of the mother
  Participants
    Vertex position | 65 | 62 | 127
    Non-vertex position | 2 | 0 | 2
Cervical dilation at labor analgesia request (cm) [Mean (Inter-Quartile Range); unit: Centimeters] — Cervical dilation at labor analgesia request (cm).Cervical dilation is measured in centimeters (cm).
  Centimeters | 3 [2 to 4] | 4 [3 to 4] | 3 [2 to 4]
VAS scores (0 to 100) at labor analgesia request [Mean (Full Range); unit: units on a scale (0 low (good)-100 high)] — VAS (verbal analogue scale) response on a 0 (no pain, good) to 100 (worst pain imaginable,bad) scale.
  units on a scale (0 low (good)-100 high) | 70 [70 to 79] | 70 [60 to 77] | 70 [60 to 79]

OUTCOME MEASURES:

1. Primary Outcome: Anesthesia Provider Administered Bolus
Description: Anesthesia provider (MD) administered boluses of additional anesthetic administered prior to the delivery of the baby.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Participants | 23 | 11

2. Secondary Outcome: VAS at 10 Centimeters Dilation of Cervix
Description: VAS (visual analogue scale) at 10 centimeters dilation of cervix on a scale of 0 (no pain,good) to 100 (worst pain imaginable,bad)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale 0 good 100 worst
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
score on a scale 0 good 100 worst | 1 [0 to 22] | 9 [0 to 36]

3. Secondary Outcome: VAS Score After Delivery
Description: VAS score (Visual Analogue Scale) on a score of 0 (no pain,good) to 100 (worst pain imaginable,bad) immediately after delivery of baby
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale 0 good-100 bad
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
score on a scale 0 good-100 bad | 0 [0 to 6] | 0 [0 to 10]

4. Secondary Outcome: Intrascapular Pain
Description: Number of participants who experienced intrascapular pain (pain in your shoulder blade) during the study period.
Time Frame: 72 hours
Measure: Number; unit: Participants
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Participants | 0 | 3

5. Secondary Outcome: Provider Administered Bolus
Description: Number of participants requiring anesthesia provider administration of additional bolus doses of pain medication.
Time Frame: 72 hours
Measure: Number; unit: participants
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
participants | 23 | 11

6. Secondary Outcome: Number of Participants Who Required Additional Provider Redoses
Description: Additional number of participants who required additional anesthesia care provider redoses of pain medication.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Participants
  0 Redoses | 44 | 51
  1 Redose | 9 | 7
  2 Redoses | 8 | 3
  3 Redoses | 5 | 1
  4 Redoses | 1 | 0

7. Secondary Outcome: Time to First Anesthesiology Provider Bolus
Description: Time elapsed in minutes from epidural set up to time to request supplemental analgesia provided by the anesthesiology care provider.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Minutes | 270 [193 to 475] | 489 [286 to 627]

8. Secondary Outcome: VAS Score Prior to First Provider Bolus Dose
Description: Patient reported visual analogue scale score (0 no pain,good-100 worst pain imaginable, bad) prior to the first anesthesiology care provider bolus dose of anesthetic (pain medication).
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale 0 good-100 bad
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
score on a scale 0 good-100 bad | 72 [50 to 82] | 61 [42 to 88]

9. Secondary Outcome: VAS Score 30 Minutes After Anesthetic Care Provider Dose
Description: Patient reported visual analogue scale score (0 no pain, good -100 worst pain imaginable, bad) 30 minutes after the first anesthesiology care provider bolus dose of anesthetic was administered to the participant for pain relief.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale 0 good-100 bad
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
score on a scale 0 good-100 bad | 25 [0 to 50] | 5 [0 to 24]

10. Secondary Outcome: Bupivacaine Consumption Per Hour
Description: Average consumption of bupivacaine in milligrams per hour.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: milligrams/hour
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
milligrams/hour | 13.1 (4) | 11.7 (3.5)

11. Secondary Outcome: Maximum Oxytocin Dose
Description: Maximum oxytocin dose administered intravenously in international units.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: International Units
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
International Units | 12 [10 to 18] | 16 [10 to 24]

12. Secondary Outcome: Time of Intrathecal Administration to Delivery
Description: Elapsed time in minutes from the intrathecal administration of anesthetic by anesthesiology provider to time of delivery of baby.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Minutes | 468 [330 to 736] | 575 [275 to 805]

13. Secondary Outcome: Number of Participants Categorized by Mode of Delivery
Description: Mode of delivery identified as: normal vaginal delivery, instrumental vaginal delivery, cesarean delivery or emergency cesarean delivery
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Participants
  Vaginal Delivery | 45 | 42
  Instrumental Delivery | 7 | 4
  Cesarean Delivery | 15 | 16

14. Secondary Outcome: PCA Boluses
Description: Number of Patient-Controlled Epidural Analgesia (PCEA) boluses of pain medication requested and number of PCEA medication boluses administered.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: Boluses
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Boluses
  Boluses Requested | 7 [4 to 13] | 8 [5 to 19]
  Boluses Delivered | 5 [3 to 9] | 5 [2 to 12]

15. Secondary Outcome: PCA Boluses Ratio
Description: The ratio of the number of Patient-Controlled Epidural Analgesia (PCEA) pain medication boluses requested and number of PCEA pain medication boluses administered by the PCEA pump.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: Ratio of requested to delivered boluses
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
Number analyzed (Participants) | 67 | 62
Ratio of requested to delivered boluses | 1.5 [1.0 to 1.7] | 1.3 [1.1 to 2.0]

ADVERSE EVENTS:
Time Frame: 72 hours after epidural catheter placement.
Description: Intrascapular pain
Arm/Group | Low Volume Bolus 0.1% Bupivacaine | High Volume Bolus .0625% Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/62
Other Adverse Events (participants affected / at risk) | 0/67 | 3/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Volume Bolus 0.1% Bupivacaine (N=67) | High Volume Bolus .0625% Bupivacaine (N=62)
Intrascapular Pain (Nervous system disorders) | 0 (0) | 3 (3) — Intrascapular pain as relating to the administration of anesthetic agents via epidural catheter.

LIMITATIONS AND CAVEATS:
A larger study would need to evaluate the secondary outcomes as the current study was underpowered to evaluate the analgesic secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03553576/Prot_SAP_000.pdf